CLINICAL TRIAL: NCT05859464
Title: A Phase I, Open-label, Multicenter Study of ZL-1218 as a Single Agent and as Combination Therapy With Anti-PD-1 Antibody to Evaluate the Safety, Tolerability, and Pharmacokinetics in Subjects With Advanced Solid Tumor Malignancies
Brief Title: A Phase 1 Study of ZL-1218 in Subjects With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Zai Lab (Hong Kong), Ltd. (Industry)
Collaborators: Zai Biopharmaceutical (Shanghai) Co., Ltd. (Unknown); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZL-1218-001; KEYNOTE-F22, MK-3475-F22 (Other: Merck Sharpe & Dohme, LLC)
Record Dates: First submitted 2023-03-17; First posted 2023-05-16 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-01

CONDITIONS: Malignant Solid Tumor
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Part 1: Dose Escalation; ZL-1218 (Experimental): Drug: ZL-1218 ZL-1218 dose escalation
  Interventions: Drug: ZL-1218
- Part 1: Dose Escalation; ZL-1218 in combination with Pembrolizumab (Experimental): Drug: ZL-1218 ZL-1218 dose escalation
  Drug: Pembrolizumab (KEYTRUDA®) Combination treatment with ZL-1218
  Interventions: Drug: ZL-1218; Drug: Pembrolizumab
- Part 2: Cohort Expansion; Prior CPI Therapy (Experimental): Drug: ZL-1218 ZL-1218 recommended dose
  Drug: Pembrolizumab (KEYTRUDA®) Combination treatment with ZL-1218
  Interventions: Drug: ZL-1218; Drug: Pembrolizumab
- Part 2: Cohort Expansion; CPI therapy Naive (Experimental): Drug: ZL-1218 ZL-1218 recommended dose
  Drug: Pembrolizumab (KEYTRUDA®) Combination treatment with ZL-1218
  Interventions: Drug: ZL-1218; Drug: Pembrolizumab

INTERVENTIONS:
Drug: ZL-1218 — ZL-1218 dose escalation
Drug: Pembrolizumab — Combination treatment with ZL-1218
  Arms: Part 1: Dose Escalation; ZL-1218 in combination with Pembrolizumab; Part 2: Cohort Expansion; CPI therapy Naive; Part 2: Cohort Expansion; Prior CPI Therapy

SUMMARY:
The purpose of this study is to characterize the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), and preliminary antitumor activity of ZL-1218 as a single agent and as combination therapy in subjects with advanced solid tumor malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Adult men and women ≥ 18 years of age. If 18 years is not the age of majority, then adult men and women ≥ age of majority per local regulation.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
* Life expectancy > 12 weeks.
* Subjects must have histologically confirmed and documented diagnosis of locally advanced unresectable or metastatic advanced solid tumor that is refractory to standard treatment, or intolerant to standard treatment, or for which no standard treatment exists.Subjects must have at least one target lesion as defined by RECIST v1.1 on CT, PET/CT, or MRI scan.
* Subjects must have a site of disease which is not previously irradiated and is safe and amenable to biopsy per the treating institution's guidelines. Subjects must be willing to undergo a tumor biopsy at screening and on treatment, per the protocol guidelines.
* Subjects must have a site of disease which is not previously irradiated and is safe and amenable to biopsy per the treating institution's guidelines. Subjects must be willing to undergo a tumor biopsy at screening and on treatment, per the protocol guidelines.

Exclusion Criteria:

* Symptomatic or uncontrolled brain metastasis requiring concurrent treatment, inclusive of but not limited to surgery, radiation, and/or corticosteroids.
* Prior exposure to CCR8 inhibitor (anti-CCR8 antibody) or hypersensitivity to any ingredient of the study drug.
* Out of range value within 10 days prior to the first dose of study treatment.
* Subjects have received a live or live-attenuated vaccine within 30 days of planned start of study therapy.
* Subjects with known history of, or any evidence of active, non-infectious pneumonitis.
* Impaired cardiac function or clinically significant cardiac disease within the last 3 months before administration of the first dose of the study drug.
* Treatment with any systemic anti-cancer treatment (including investigational products) within 4 weeks before first dose of study drug.
* Non-palliative radiotherapy within 2 weeks prior to first dose of study drug or have had history of radiation pneumonitis.
* Major surgery within 4 weeks of the first dose of study drug.
* Infections requiring systemic antibiotic therapy.
* Any medical conditions that would, in the investigator's judgement, prevent the subject's participation in the clinical study due to safety concerns, compliance with the study procedures, or interpretation of the study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2023-07-24 (Actual); Primary Completion 2025-08-28 (Actual); Study Completion 2025-08-28 (Actual)

PRIMARY OUTCOMES:
Incidence of Dose Limiting Toxicities | Approximately 24 months
  Number of subjects with dose limiting toxicities (DLTs) through dose escalation only.
Incidence of Treatment Emergent Adverse Events | Approximately 24 months
  Number of subjects with treatment-emergent adverse effects through dose escalation and expansion.
Incidence of Serious adverse events | Approximately 24 months
  Number of subjects with Serious Adverse Events through dose escalation and expansion.
Clinically Significant changes in safety assessments | Approximately 24 months
  Changes in safety assessment parameters (e.g., vital signs, electrocardiograms [ECGs], and clinical laboratory results) through dose escalation and expansion.
ORR per RECIST 1.1 | up to 24 months
  Objective Response Rate (ORR) per RECIST 1.1 through dose expansion only.
ORR per iRECIST | up to 24 months
  Objective Response Rate per iRECIST through dose expansion only.

SECONDARY OUTCOMES:
ORR per RECIST 1.1 | up to 24 months
  Objective Response Rate (ORR) per RECIST 1.1 through dose escalation only.
ORR per iRECIST | up to 24 months
  Objective Response Rate (ORR) per iRECIST through dose escalation only.
Duration of Response per RECIST 1.1 | up to 24 months
  Duration of Response per RECIST 1.1 through dose escalation and expansion.
Duration of Response per iRECIST | up to 24 months
  Duration of Response per iRECIST through dose escalation and expansion.
PFS per RECIST 1.1 | up to 24 months
  Progression-Free Survival (PFS) per RECIST 1.1 through dose escalation and expansion.
PFS per iRECIST | up to 24 months
  Progression-Free Survival (PFS) per iRECIST through dose escalation and expansion.
DCR per RECIST 1.1 | up to 24 months
  Disease Control Rate (DCR) per RECIST 1.1 through dose escalation and expansion.
DCR per iRECIST | up to 24 months
  Disease Control Rate (DCR) per iRECIST through dose escalation and expansion.
Overall Survival | up to 24 months
  Overall Survival (OS) through dose escalation and expansion.
Pharmacokinetics (PK): AUC | up to 24 months
  Area under curve (AUC) through dose escalation and expansion.
Pharmacokinetics (PK): Cmax | up to 24 months
  Maximum serum concentration (CMax) through dose escalation and expansion.
Pharmacokinetics (PK): Tmax | up to 24 months
  Time to reach Cmax (Tmax) through dose escalation and expansion.
Pharmacokinetics (PK): Ctrough | up to 24 months
  Ctrough through dose escalation and expansion.
Pharmacokinetics (PK): Vss | up to 24 months
  Volume of distribution as steady state (Vss) through dose escalation and expansion.
Pharmacokinetics (PK): CL | up to 24 months
  Clearance (CL) through dose escalation and expansion.
Pharmacokinetics (PK): t1/2 | up to 24 months
  Half-life (t1/2) through dose escalation and expansion.
Immunogenicity | up to 24 months
  Incidence of anti-drug antibodies (ADAs) through dose escalation and expansion.
Immunogenicity | up to 24 months
  Quantity of anti-drug antibodies (ADAs) through dose escalation and expansion.

CONTACTS AND LOCATIONS:
Locations (15):
- United States (5):
  - Zai Lab Site 2005, Irvine, California
  - Zai Lab Site 2007, Detroit, Michigan
  - Zai Lab Site 2001, Hackensack, New Jersey
  - Zai Lab Site 2002, New York, New York
  - Zai Lab Site 2003, Spokane, Washington
- China (2):
  - Zai Lab Site 1002, Hangzhou
  - Zai Lab Site 1001, Shanghai
- Spain (8):
  - Zai Lab Site 8005, Barcelona, Barcelona
  - Zai Lab Site 8001, Barcelona, Barcelona
  - Zai Lab Site 8007, Madrid, Madrid
  - Zai Lab Site 8008, Madrid, Madrid
  - Zai Lab Site 8004, Pozuelo de Alarcón, Madrid
  - Zai Lab Site 8003, Seville, Sevilla
  - Zai Lab Site 8002, Valencia, Valencia
  - Zai Lab Site 8006, Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No